CLINICAL TRIAL: NCT04431817
Title: Operational Analysis of Depth Camera to Assist Gait Analysis in Outpatient Rehabilitation for Unilateral Transtibial and Transfemoral Amputees
Brief Title: KinetiGait- Analysis of Depth Camera to Assist Gait Analysis for Unilateral Transtibial/Transfemoral Amputees
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 189608
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Lower Limb Amputation
Keywords: depth camera, gait analysis, LE loss, SMs and Veterans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Left transtibial: Left below knee amputation- 25
  Interventions: Device: KinetiGait
- Right transtibial: Right below knee amputation- 25
  Interventions: Device: KinetiGait
- Left transfemoral: Left above knee amputation- 25
  Interventions: Device: KinetiGait
- Right transfemoral: Right above knee amputation- 25
  Interventions: Device: KinetiGait
- Provider: Provider- 15
  Interventions: Device: KinetiGait

INTERVENTIONS:
Device: KinetiGait — This device is an Intel RGB depth camera that relays video to gait analysis software. The images will be taken from amputees walking at a self-selected pace on a treadmill.

SUMMARY:
This is a feasibility study about implementing and using the KinetiGait gait analysis system in clinical practice to enhance the rehabilitation of service members with lower limb disfunction. There will be questionnaires completed by participants and surveys completed by both participant and provider.

DETAILED DESCRIPTION:
We propose a feasibility study about implementing and using the KinetiGait gait analysis system in clinical practice to enhance the rehabilitation of service members with lower limb dysfunction. Up to 100 subjects will be consented, with the expectation that 80% (e.g., n=80) will complete the study with a complete dataset. Baseline sessions will consist of 7 minutes of walking at a self-selected speed between 0.7 and 1.3 m/s, after which participants will take the PLUS-M 12 Item Short Form and PROMIS-29 questionnaires, as well as a short survey. Participants will complete the questionnaires again at 1 month and 3 month. Providers who observed/operated the KinetiGait system will also take a short survey on ease of use and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral or transtibial amputee
* Fitted by a prosthetist at a Military Treatment Facility
* K2-K4 Medicare Functional Classification Levels
* DEERS-eligible.
* For providers: MHS provider

Exclusion Criteria:

* K0-K1 Medicare Functional Classification Levels
* Physically unstable or requires an ambulatory device
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include individuals who are DEERS-eligible between the ages of 18 and 65 and in K2-K4 Medical Functional Classification levels. The providers must be MHS providers.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Prosthetic Limb Users Survey of Mobility (PLUS-M) | 5-10 minutes
  12-item short form to assess functional status, quality of life and perceived mobility.
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 | 5-10 minutes
  Measures self-reported capability rather than actual performance of physical capabilities.

SECONDARY OUTCOMES:
Provider survey | 5-10 minutes
  Survey for providers indicating age, level of clinical training, experience with gait analysis and views on integrating technology into the clinical environment.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel M Kim, M.D., Principal Investigator — WRNMMC
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273